CLINICAL TRIAL: NCT02126631
Title: Comparison of a Sternal ECG Patch With a Standard Recording System for Holter Monitoring
Brief Title: Sternal ECG Patch Comparison Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bardy Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 6147
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Syncope; Presyncope; Palpitations; Atrial Fibrillation; Supraventricular Tachycardia
MeSH Terms: conditions — Syncope; Atrial Fibrillation; Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is intended to compare the new Carnation Ambulatory Monitoring (CAM) System, a patch monitoring system, with the Holter monitoring system. Holters represent the current standard for continuous recording of the ECG over extended periods.

DETAILED DESCRIPTION:
The purpose of this research is to simplify the system of recording ECGs. Carnation Ambulatory Monitoring (CAM) System is a small patch system that can be worn during most activities include showering. Each patient will be his or her own control, and will wear the CAM and Holter systems simultaneously for 24 hours. Both systems will then be sent out for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Syncope of uncertain etiology or
* Pre-syncope of uncertain etiology or
* Palpitations of uncertain etiology or
* Management of known AF/SVT patients

Exclusion Criteria:

* Any dermatitis or infected skin over the sternum (Carnation patch) or left upper anterior thorax (Zio patch).
* A sternal or thoracic incision that extends under the patch within 3 months from the date of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac patients at Auckland City Hospital, Auckland, New Zealand
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
ECG signal quality | 24 hours of patient use, plus shipping and analysis time ~ 2 weeks
  ECG signal quality = scoring the ability of each system to record electrical activity from the atrium (P-waves). The Physician Event Committee will independently score the P-waves from all recordings, using the following scale: Excellent, Good, Fair, Poor, Non-existent. Diagnostic yield will also be assessed.

SECONDARY OUTCOMES:
Device comfort | 24 hours
  Secondary outcome measures will include Human Factors performance of the 2 systems, which will be scored and compared in the following areas and duration of patch adherence: skin irritation, comfort, contact and stability.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Hunt, PhD, Study Director — Bardy Diagnostics, Inc. (sponsor); Warren Smith, MBChB, Principal Investigator — Auckland City Hospital
Locations (1):
- Auckland City Hospital, Auckland, New Zealand